CLINICAL TRIAL: NCT01368328
Title: Effect of Chromium Supplementation on Insulin Sensitivity in Patients With Type 2 Diabetes
Brief Title: Effect of the Chromium Nicotinate on Type 2 Diabetes
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidade Federal de Goias (Other)
Responsible Party: Marília Mendonça Guimarães, Faculdade de Nutrição Universidade Federal de Goiás
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DM2
Record Dates: First submitted 2011-04-12; First posted 2011-06-07 (Estimated); Last update posted 2011-06-07 (Estimated); Status verified 2011-02

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 Diabetes; Chromium; Insulin resistance
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance | interventions — chromium nicotinic acid complex

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Chromium nicotinate
- Chromium nicotinate 50 mcg (Active Comparator)
  Interventions: Dietary Supplement: Chromium nicotinate
- Chromium nicotinate 200 mcg (Active Comparator)
  Interventions: Dietary Supplement: Chromium nicotinate

INTERVENTIONS:
Dietary Supplement: Chromium nicotinate — The intervention is offered during three months. There is a placebo group, chromium nicotinate 50 mcg group and chromium nicotinate 200 mcg group. Each patient is oriented to consume one capsule one hour after lunch and one capsule one hour after dinner.

SUMMARY:
The role of micronutrients in diabetes is not well understood. Studies have demonstrated the relationship between low chromium serum levels and insulin resistance. This study aims to evaluate the effect of chromium nicotinate on increasing insulin sensitivity in patients with type 2 diabetes.

DETAILED DESCRIPTION:
Insulin is a hormone secreted by cells β of pancreatic islets in response to increased levels of glucose and serum amino acids. Insulin resistance means a decrease in the ability of insulin to stimulate glucose utilization because is disabled in the insulin receptor, decrease in concentration of receptors or failure mechanism of cell transit. Recently, the discovery of a substance called low molecular weight chromium-binding substance (LMWCr), showed the ability of this substance in amplifying insulin signaling, increasing the sensitivity of insulin receptors in the plasma membrane. This way, the capacity of LMWCr in activating the insulin receptor depends on levels of serum chromium. Thus, the hypothesis that the nutritional status of individual poor chromium contributes to the decrease in glucose tolerance and consequently, for type 2 Diabetes. Thus, it becomes necessary to assess the effect of supplementation of chromium in increased insulin sensitivity in patients with type 2 Diabetes. This is a double-blind randomized clinical trial, consisting of a period of three months of nutritional intervention with chromium nicotinate, biochemical and anthropometric evaluation and assessment of food profile and physical activity.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Body mass index > 25 kg/m2
* Increased waist circumference

Exclusion Criteria:

* Subjects on insulin
* Pregnancy
* Patients with chronic complications as heart disease, nephropathy, retinopathy

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 57 (Estimated)
Dates: Start 2010-03; Primary Completion 2011-07 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
Insulin Sensitivity as assessed with homeostatic model assessment (HOMA) | baseline, 45 days and 90 days

SECONDARY OUTCOMES:
fasting triglycerides, high density lipoprotein cholesterol, low density lipoprotein cholesterol | baseline, 45 days and 90 days
body weight | baseline, 45 days, 90 days
body fat accessed with bioimpedance | baseline, 45 days, 90 days
waist circumference | baseline, 45 days, 90 days
urea and creatinine | baseline, 45 days, 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Marília Mendonça Guimarães, Principal Investigator — Faculdade de Nutrição - Universidade Federal de Goiás; Maria Sebastiana Silva, Principal Investigator — Faculdade de Educação Física - Universidade Federal de Goiás
Locations (1):
- Goiania Municipal Health Departament, Goiânia, Goiás, Brazil

REFERENCES:
- [Background] Anderson RA. Chromium and insulin resistance. Nutr Res Rev. 2003 Dec;16(2):267-75. doi: 10.1079/NRR200366. PMID 19087394
- [Background] Kleefstra N, Houweling ST, Bakker SJ, Verhoeven S, Gans RO, Meyboom-de Jong B, Bilo HJ. Chromium treatment has no effect in patients with type 2 diabetes in a Western population: a randomized, double-blind, placebo-controlled trial. Diabetes Care. 2007 May;30(5):1092-6. doi: 10.2337/dc06-2192. Epub 2007 Feb 15. PMID 17303791
- [Background] Kleefstra N, Houweling ST, Jansman FG, Groenier KH, Gans RO, Meyboom-de Jong B, Bakker SJ, Bilo HJ. Chromium treatment has no effect in patients with poorly controlled, insulin-treated type 2 diabetes in an obese Western population: a randomized, double-blind, placebo-controlled trial. Diabetes Care. 2006 Mar;29(3):521-5. doi: 10.2337/diacare.29.03.06.dc05-1453. PMID 16505499
- [Background] Martin J, Wang ZQ, Zhang XH, Wachtel D, Volaufova J, Matthews DE, Cefalu WT. Chromium picolinate supplementation attenuates body weight gain and increases insulin sensitivity in subjects with type 2 diabetes. Diabetes Care. 2006 Aug;29(8):1826-32. doi: 10.2337/dc06-0254. PMID 16873787
- [Background] Ghosh D, Bhattacharya B, Mukherjee B, Manna B, Sinha M, Chowdhury J, Chowdhury S. Role of chromium supplementation in Indians with type 2 diabetes mellitus. J Nutr Biochem. 2002 Nov;13(11):690-697. doi: 10.1016/s0955-2863(02)00220-6. PMID 12550067
- See also: American Diabetes Association — http://www.diabetes.org/